CLINICAL TRIAL: NCT01462838
Title: Phase I/IIa Study of Immunization With a p16INK4a Peptide Combined With MONTANIDE ISA-51 VG in Patients With Advanced HPV-associated Cancers
Brief Title: Immune Therapy of HPV-induced Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oryx GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VicOryx
Record Dates: First submitted 2011-10-25; First posted 2011-10-31 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: HPV-induced Cancers
Keywords: advanced HPV-; p16INK4a-positive; cervical; vulvar,; vaginal; penile; anal; head; neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunization (Experimental): P16_37-63 peptide plus Montanide ISA-51 VG
  Interventions: Biological: P16_37-63

INTERVENTIONS:
Biological: P16_37-63 — 100 ug per application subcutaneously, mixed with 0.3 ml Montanide ISA-51 VG; once a week for four weeks, followed by a 4 week rest period (1 cycle), up to 3 cycles

SUMMARY:
Patients with advanced HPV- and p16INK4a-positive cancers will receive the peptide P16_37-63 in combination with Montanide® ISA-51 VG so that an immune response directed against the tumor cells can be induced. The aim is to show that vaccination with P16_37-63 is safe and can induce or enhance immune responses against p16INK4a.

DETAILED DESCRIPTION:
The present study is initiated to evaluate vaccination with P16_37-63 -peptide in patients with advanced HPV- and p16INK4a -positive cervical, vulvar, vaginal, penile, anal or head and neck cancer. Specifically, the present study aims at the following questions:

* Evaluation of potential toxicity of the vaccination with P16_37-63 -peptide
* Evaluation of the immune response in patients with advanced HPV- and p16INK4a-positive cervical, vulvar, vaginal, penile, anal or head and neck cancer before vaccination and after vaccination with P16_37-63.

In this context, the present study shall demonstrate whether application of P16_37-63 in a vaccination approach is associated with the induction of peptide-related toxicity. Hence, the study marks the first step towards the application of P16_37-63 in humans, as it provides information on the safety of P16_37-63 as vaccination agent for the first time. Moreover, the study shall provide initial information, whether vaccination with P16_37-63 can induce p16INK4a -specific immune responses in patients with advanced HPV- and p16INK4a -positive cervical, vulvar, vaginal, penile, anal or head and neck cancer. Thus, it shall provide information, whether P16_37-63 has the potential to elicit peptide-specific immune responses and therefore represent a suitable target for the induction of tumor antigen-specific immune responses in this population.

The present study marks an important milestone towards a potential application of P16_37-63 as therapeutic agent in the management of patients with advanced HPV- and p16INK4a -positive cervical, vulvar, vaginal, penile, anal or head and neck cancer. Long-term goal of this approach is to develop novel tools for the palliative and/or adjuvant therapy of patients with advanced advanced HPV- and p16INK4a -positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, advanced HPV-positive cervical, vulvar, vaginal, penile, anal or head and neck cancer cancers under progression, regression or with stable disease after standard therapy (and still incurable) or after refusal of standard therapy or with contraindications for standard treatment
* HPV positivity as tested by HPV genotyping from paraffin embedded tumor tissue
* Diffuse expression of p16INK4a in the tumor as analyzed by immunohistochemistry on paraffin embedded tumor tissue.
* Expected survival of at least six months.
* Full recovery from surgery, chemo therapy or radiation therapy.
* ECOG performance status 0, 1 or 2.
* The following laboratory results:

Neutrophil count ≥ 1.5 x 109/L Lymphocyte count ≥ 0.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin < 2mg/dL

* Male or female patients ≥ 18 years old
* Patient´s written informed consent for participation in the trial

Exclusion Criteria:

* Prior treatment with P16_37-63 peptide
* Clinically significant heart disease (NYHA Class III or IV).
* Other serious illnesses, eg, serious infections requiring antibiotics or bleeding disorders.
* History of immunodeficiency disease or autoimmune disease.
* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available.
* HBV, HCV or HIV positivity.
* Chemotherapy, any type of radiation therapy, or immunotherapy within 4 weeks before study entry
* Concomitant treatment with steroids, antihistaminic drugs, or nonsteroidal anti-inflammatory drugs (unless used in low doses for prevention of an acute cardiovascular event or for pain control). Topical or inhalational steroids are permitted.
* Participation in any other clinical trial involving another investigational agent within 4 weeks.
* Pregnancy or lactation.
* Women of childbearing potential who are not using a medically acceptable means of contraception.
* Psychiatric or addictive disorders that may compromise the ability to give informed consent.
* Lack of availability of a patient for immunological and clinical follow-up assessment.
* Brain metastases (symptomatic and non-symptomatic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Immune response | every 2 weeks
  Immune response against peptide P16_37-63. A positive immune response is defined as positive DTH response against peptide P16_37-63 or a humoral (ELISA for the detection of p16-specific IgG/IgM/IgA) and/or CD8 and/or CD4 cellular (IFN gamma ELISpot for the detection of p16INK4a-specific T cells) immune response exceeding the assay specific cut-off values for a positive response against peptide P16_37-63.

SECONDARY OUTCOMES:
Tumor response | every 8 weeks
  assessed by CT or MRI scans according to RECIST
safety | up to 8 months
  number and severity of adverse events categorized according to CTC criteria version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jäger, Prof. Dr., Principal Investigator — Krankenhaus Nordwest Frankfurt
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany